CLINICAL TRIAL: NCT02460055
Title: Randomized Controlled Trial Examining Effect Of Endotracheal Tube Intubation On Dysphagia In Children Presenting For Upper GI Endoscopy
Brief Title: Trial- Dysphagia From ETT or GI Endoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no subject met enrollment criteria
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Imelda Michelle Tjia, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-32691
Record Dates: First submitted 2015-02-27; First posted 2015-06-02 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Dysphagia; Respiratory Complications
Keywords: EGD Dysphagia; ETT Intubation dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Propofol; Fentanyl; Dexamethasone; Ondansetron; Sevoflurane; Nitrous Oxide; Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endotracheal tube (Active Comparator): Following routine inhalation induction with 8% sevoflurane in oxygen and nitrous oxide, 100% oxygen will be administered and intravenous access will be secured. Intravenous administration of Propofol 3mg/kg and Fentanyl 1mcg/kg will be administered to facilitate endotracheal intubation with an age appropriate endotracheal tube. Presence of an audible air leak around the endotracheal tube will be addressed by inflating the cuff with air until the audible leak is no longer appreciated. The endotracheal tube will not be lubricated prior to intubation. Other medications that will be administered during the procedure include Dexamethasone at a dose of 0.15mg/kg up to 20 mg and Ondansetron 0.15mg/kg up to 4mg.
  Interventions: Device: endotracheal tube; Drug: propofol; Drug: Fentanyl; Drug: Dexamethasone; Drug: Ondansetron; Drug: sevoflurane, nitrous oxide and oxygen
- No Endotracheal tube (Active Comparator): Those not receiving endotracheal intubation will undergo an inhalation induction, have intravenous access secured and intravenous propofol 3mg/kg with Fentanyl 1mcg/kg will be administered prior to placement of the nasal trumpet and connection to the anesthesia circuit.patients will receive a general anesthetic consisting of sevoflurane in oxygen and air at routine concentrations for maintenance of anesthesiaOther medications that will be administered during the procedure to both arms of patients include Dexamethasone which will be administered at a dose of 0.15mg/kg up to 20 mg and Ondansetron 0.15mg/kg up to 4mg for post operative nausea and vomiting prophylaxis.
  Interventions: Drug: propofol; Drug: Fentanyl; Drug: Dexamethasone; Drug: Ondansetron; Drug: sevoflurane, nitrous oxide and oxygen

INTERVENTIONS:
Device: endotracheal tube — This study will determine if the placement of an ETT will lead to dysphagia.
  Arms: Endotracheal tube
Drug: propofol — propofol 3mg/kg will be administered to facilitate endotracheal intubation
Drug: Fentanyl — Fentanyl 1mcg/kg will be administered to facilitate endotracheal intubation
Drug: Dexamethasone — Dexamethasone 0.15mg/kg up to 20 mg will be used for anti-emesis prophylaxis
Drug: Ondansetron — Ondansetron 0.15mg/kg up to 4mg will be used for anti-emesis prophylaxis
Drug: sevoflurane, nitrous oxide and oxygen — Inhalational agents will be used to induce general anesthesia

SUMMARY:
The purpose of this study is to conduct a randomized clinical trial to compare the incidence of dysphagia in patients receiving general anesthesia with and without an endotracheal tube for Upper gastrointestinal endoscopy. If the incidence of dysphagia is found to be increased following endotracheal intubation for this procedure it could influence the investigators practice as anesthesiologists and may mandate the future routine use of laryngeal tracheal application of lidocaine at the time of intubation for example.

DETAILED DESCRIPTION:
Patients between the ages of 5-17 with normal cognitive function presenting for Upper GI endoscopy will be considered for participation in this study. After consent is obtained from the parent/legal guardian, the patient will undergo a general anesthetic to facilitate the procedure. All patients in this study will receive a general anesthetic. Following routine inhalation induction with 8% sevoflurane in oxygen and nitrous oxide, 100% oxygen will be administered and intravenous access will be secured. Intravenous administration of Propofol 3mg/kg and Fentanyl 1mcg/kg will be administered to facilitate endotracheal intubation with an age appropriate endotracheal tube for children randomized to receive endotracheal intubation. Following endotracheal intubation, the oropharynx will be auscultated for the presence of an audible air leak around the endotracheal tube. If an audible leak is appreciated below 20cm of H2O pressure, the cuff of the endotracheal tube will be gradually inflated with air until the audible leak is no longer appreciated. This is routine practice following endotracheal intubation. The endotracheal tube will not be lubricated prior to intubation. Those not receiving endotracheal intubation will undergo an inhalation induction, have intravenous access secured and intravenous propofol 3mg/kg with Fentanyl 1mcg/kg will be administered prior to placement of the nasal trumpet and connection to the anesthesia circuit. Both arms of patients will receive a general anesthetic consisting of sevoflurane in oxygen and air at routine concentrations for maintenance of anesthesia either via the endotracheal tube or via nasal trumpet for the Upper GI endoscopy procedure. Other medications that will be administered during the procedure to both arms of patients include Dexamethasone which will be administered at a dose of 0.15mg/kg up to 20 mg and Ondansetron 0.15mg/kg up to 4mg for post operative nausea and vomiting prophylaxis. Additional maneuvers which may aggravate post operative dysphagia such as the use of a Yankauer suction catheters, placement of nasopharyngeal temperature probes and coughing during emergence prior to extubation of the patient will be avoided. Utilization of soft tip suction catheters and skin or axilla temperature probes will be employed and the trachea will be extubated under deep anesthesia. Data that will be collected will include: Pre-operative data: the recent need of breathing treatments, allergy history and smokers at home. Intraoperative data: the presence of bucking/coughing during intubation, experience level of the intubating practitioner, laryngoscopic view, endotracheal tube size, number of intubation attempts, experience of the endoscopist, size of the endoscope used and duration of the procedure. With both techniques (intubation and nasal trumpet use), the data that will be collected will include: Coughing or bucking prior to extubation or during emergence and removal of nasal trumpet, occurence of laryngospasm, bronchospasm or desaturation less than 95% requiring treatment , breath-holding and methods for resolution. PACU data: Incidence of laryngospasm, breath-holding, or apnea, presence or absence of nausea/vomiting and if treatment was required, requirement of additional pain medication, documentation of dysphagia prior to the first oral intake and grading of the sore throat as previously documented. Postoperatively, the presence of dysphagia will be sought at two different time points: Via face to face interview in the post operative anesthesia care unit (PACU) prior to the first per oral intake and 24 hours later at which point presence/absence of dysphagia will be ascertained via phone. Complaints will be graded according to a scoring system (Capon LM et al. Anesthesiology 1983) : Presence of sore throat (ST): Yes/No If No, ST will be graded as 0= no sore throat If Yes, ST will be graded 1-3 as follows: 1=mild sore throat (pain with swallowing) 2=moderate sore throat (pain present constantly and worsens with swallowing) 3=severe sore throat (pain interferes with eating and requires analgesic medication for relief). Pain will also be assessed with a VAS score immediately postoperatively and at 24 hours

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 5-17 with normal cognitive function, without medical comorbidities who are scheduled to undergo esophagogastroduodenoscopy under general anesthesia will be recruited for the study

Exclusion Criteria:

* Patients under the age of five, or those between ages 5-17 years with cognitive delay or neurological disease scheduled to undergo Upper GI endoscopy will be excluded.
* Patients who currently have a sore throat or had a sore throat within the past one week will not be included in this study.
* Other patients with cardiopulmonary disease, coagulopathies, hepatorenal disease, endocrinological disease or airway abnormalities will also be excluded.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Dysphagia | up to 24 hours
  Dysphagia will be determined by a scale ( 0=no sore throat, 1=mild sore throat, 2=moderate sore throat, 3=severe sore throat) and Visual analog scale .

SECONDARY OUTCOMES:
Patient Satisfaction | up to 24 hours
  Patient satisfaction will be measured by a patient satisfaction survey prior to discharge from PACU

OTHER OUTCOMES:
Time efficiency with no ETT Intubation | up to 24 hours
  Efficiency will be measured by OR times between patients.
Respiratory Compromise | up to 24 hours
  Data will be collected for different phases of anesthesia care for episodes of desaturation, laryngospasm, apnea, coughing: induction, intraoperatively and postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Imelda M Tjia, MD, Principal Investigator — Baylor College of Medicine

IPD SHARING:
Plan to Share IPD: Undecided